CLINICAL TRIAL: NCT05209828
Title: Prospective, Monocentric Observational Study on the Clinical Use and Patient Satisfaction of Pfmmedical Implantable Vascular Access Ports
Brief Title: Post-market Clinical Follow-up of Pfmmedical Ports
Status: Completed | Type: Observational
Sponsor: pfm medical gmbh (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF study pfmmedical Ports
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-11

CONDITIONS: Vascular Access Port; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- pfmmedical port implantation: Port implantation for continous vascular access.
  Interventions: Device: pfmmedical implantable vascular access ports

INTERVENTIONS:
Device: pfmmedical implantable vascular access ports — Implantion of an implantable vascular access port which facilitates repeated vascular access intended for the delivery of medications, intravenous fluids, parenteral nutrition solutions or blood products and blood sampling using a Huber needle.
  Other Names: Jet Port® Plus II Contrast; T-Port Contrast; T-Port Low Profile Contrast

SUMMARY:
Prospective, monocentric, non-randomised, observational post-market clinical follow-up study in Germany to obtain post-market information on the pfmmedical ports with a follow-up (FU) of 6 months. The focus is on patient reported satisfaction, clinical application, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years.
* Medical indication for port catheter implantation.
* The patient is mentally able to understand the nature, aims and possible consequences of the PMCF study.
* Patient information has been provided and written consent exists.

Exclusion Criteria:

* Contraindications according to the manufacturer´s instructions for use (IFU).
* The patient is institutionalised by court or official order (MPDG §27).
* Patient participates in another operative clinical investigation if it relates to the area of port devices and/or influences the primary endpoint of the PMCF study.
* Patients who currently already have a port implanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients requiring repeated vascular access
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Patients satisfaction | 6 months after port implantation
  The study hypothesis is that the patients' satisfaction after the study intervention is not worse than the satisfaction identified in the current literature. Satisfaction is determined using the patient questionnaire (6 months after implantation).
  The following 4 domains of the validated questionnaire by Nagel et.al., 2012 are considered as relevant for the clinical outcome:
  * Overall, how satisfied are you with the port system?
  * In a similar situation, would you choose the port again?
  * How satisfied are you with the cosmetic result?
  * Does the port cause pain?

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Knebel, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagel SN, Teichgraber UK, Kausche S, Lehmann A. Satisfaction and quality of life: a survey-based assessment in patients with a totally implantable venous port system. Eur J Cancer Care (Engl). 2012 Mar;21(2):197-204. doi: 10.1111/j.1365-2354.2011.01275.x. Epub 2011 Aug 18. PMID 21851433
- See also: manufacturer homepage of the investigational devices — https://www.pfmmedical.com/productcatalogue/2051/index.html